CLINICAL TRIAL: NCT03650491
Title: A Phase I Study of FOR46 Administered Every 21 Days in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: A Study of FOR46 in Patients With Relapsed or Refractory Multiple Myeloma (RRMM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fortis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FOR46-002
Record Dates: First submitted 2018-08-21; First posted 2018-08-28 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma With Failed Remission
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Following completion of the dose escalation phase of the study and determination of a recommended phase 2 dose, patients will be enrolled into a dose expansion cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: FOR46 (Dose Escalation) (Experimental): Eligible patients will receive FOR46 administered as an IV infusion every 21 days. Patients will be enrolled into escalating dose levels during the Dose Escalation period of the study.
  Interventions: Drug: FOR46
- Experimental: FOR46 (Dose Expansion) (Experimental): Eligible patients will receive FOR46 administered as an IV infusion every 21 days. Patients will receive the maximum tolerated dose during the Dose Expansion period of the study.
  Interventions: Drug: FOR46

INTERVENTIONS:
Drug: FOR46 — FOR46 is an intravenously (IV) administered antibody-drug conjugate (ADC) directed against CD46

SUMMARY:
This study will test the safety and efficacy of FOR46 given every 21 days to patients with relapsed or refractory multiple myeloma.

The name of the study drug involved in this study is: FOR46 for Injection

DETAILED DESCRIPTION:
This study is designed to evaluate the safety, tolerability and antitumor activity of FOR46 in patients with relapsed or refractory multiple myeloma. This study will be conducted in two parts:

Dose escalation:

This part will evaluate increasing doses of FOR46 to identify the maximum tolerated dose (MTD). The first patient enrolled on the study will receive the lowest dose of FOR46. Once this dose is shown to be safe, a second patient will be enrolled at the next higher dose. Patients will continue to be enrolled into either single or multiple patient groups receiving increasing doses until the MTD is reached.

Dose expansion:

This part of the study will further evaluate the safety, tolerability and antitumor activity of FOR46 at a dose shown to be safe in the dose escalation part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Measurable MM that is relapsed or refractory to established therapies with known clinical benefit in RRMM or intolerant of those established MM therapies. Prior lines of therapy must include a proteasome inhibitor (PI), an immunomodulatory imide drug (IMiD) and a CD38-directed therapy in any order of combination.
* ECOG performance status of 0 or 1
* Adequate hematologic, renal and hepatic function
* Females of child-bearing potential must have a negative serum pregnancy test and use a medically acceptable form of contraception
* Male patients with with female partners of childbearing potential must agree to use 2 effective methods of contraception
* Patients must provide signed informed consent

Exclusion Criteria:

* Persistent clinically significant toxicities from previous anticancer therapy
* NCI CTCAE Grade ≥ 2 peripheral neuropathy from any etiology or has a genetic disorder that is associated with peripheral neuropathy even without current neuropathic manifestations
* Has received treatment with a stem cell transplant within 12 weeks before administration of patient's first dose of FOR46
* Has had radiation or systemic anticancer therapy within 14 days before first dose of FOR46
* Has received treatment with an investigational drug within 28 days before first dose of FOR46
* Has had a major surgical procedure within 28 days before administration of the patient's first FOR46 dose
* Is breastfeeding
* Clinically significant cardiovascular disease
* Uncontrolled, clinically significant pulmonary disease
* Uncontrolled intercurrent illness
* Has known positive status for HIV or either active/chronic hepatitis B/C
* Requires anticoagulation with warfarin or direct thrombin inhibitor; a washout of 7 days before the administration of a patient's first FOR46 dose is required for patients removed from these treatments
* Requires medications that are strong inhibitors or strong inducers of CYP3A4
* Has a history of episodic atrial fibrillation or flutter; patients with chronic atrial fibrillation are not excluded.
* Prior treatment with an ADC containing Monomethyl auristatin E (MMAE) or Monomethyl auristatin F (MMAF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Through 1 month following last dose
  Number of patients with treatment-related adverse events as assessed by NCI CTCAE v5.0.
Occurrence of dose-limiting toxicities | Through 1 month following last dose
  The severity and incidence of dose-limiting toxicities related to escalating dose levels of FOR46
Disease response | 6 months
  Overall response rate of FOR46, defined as all responses greater than or equal to a partial response, complete response, stringent complete response, or minimal residual disease negativity

SECONDARY OUTCOMES:
Characterize FOR46 plasma concentration | Through 1 month following last dose
  FOR46 maximum plasma concentration
Characterize the FOR46 area under the curve | Through 1 month following last dose
  FOR46 area under the plasma concentration-time curve
Characterize FOR46 elimination | Through 1 month following last dose
  FOR46 elimination half-life
Antidrug Antibodies | Through 1 month following last dose
  Change from baseline in serum levels of antidrug antibodies
Duration of response | From first dose through 6 months following last dose
  Assessed by IMWG criteria
Progression-free survival | From first dose through 6 months following last dose
  Assessed by IMWG criteria
Time to progression | From first dose through 6 months following last dose
  Assessed by IMWG criteria

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dorr, MD, Study Director — Fortis Therapeutics, Inc.
Locations (7):
- United States (7):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center, Johns Hopkins University, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University in St. Louis-Siteman Cancer Center, St Louis, Missouri
  - Icahn School of Medicine at Mt. Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No